CLINICAL TRIAL: NCT04637854
Title: Posture Analysis During Dental Surgery Using Visual Markers: a Randomized Controlled Clinical Trial (RCT)
Brief Title: Postural Analysis During Dental Surgery
Acronym: PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Giovanni Lodi, Associate Professor, University of Milan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PAD
Record Dates: First submitted 2020-11-10; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Postural Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Operating Microscope. (Experimental): Surgical technique is the same used for extraction of the lower third molar. Patients will be enrolled (baseline) whenever sign their written informed consent to participate to the study, after having read and understand the informative pamphlet.
  The intervention will be performed under local anesthesia (mepivacaine 20 mg/ml with adrenaline 1:100000) and by the use of microscope.
  At the end of the surgical procedure, all patients will receive a 100mg Nimesulide cpr and apply the ice pack on the cheek.
  At the end of each procedure will give post-operative instructions for all patients and prescribe an antiseptic therapy with chlorhexidine coll. 0.2% 3 times/ day for 10 days from the day following the intervention and anti-inflammatory therapy Nimesulide 100 mg cpr to take up to 2 times / day for up to 4 days.
  Each patients will be recalled for follow-up visits at 7 days.
  Interventions: Procedure: Operating microscope
- Surgical Loupes with coaxial illumination. (Active Comparator): The same as above but the intervention will be performed with the use of surgical loupes
  Interventions: Procedure: Surgical loupes
- Naked Eye. (Active Comparator): The same as above but the intervention will be performed at naked eyes
  Interventions: Procedure: Naked eyes

INTERVENTIONS:
Procedure: Operating microscope — Third molar extraction using microscope
  Arms: Operating Microscope.
Procedure: Surgical loupes — Third molar extraction using loupes with co-axial illumination
  Arms: Surgical Loupes with coaxial illumination.
Procedure: Naked eyes — Third molar extraction using naked eyes
  Arms: Naked Eye.

SUMMARY:
Background: Attention and awareness towards MSDs in the dental profession has increased considerably in recent years. From recent literature reviews, it is learned that prevalence of MSDs in dentists is 64-93%. It has been seen that the use of magnification systems not only improves the operator's visual capabilities, but also allows for a more correct posture, and to prevent the onset of back and neck disorders.

Purpose and methods: Evaluate dentist posture during extraction of third lower molars depending on whether the operator uses the naked eye, surgical loupes or surgical microscope systems. Data will be evaluated through the index RULA (rapid upper limb assesment) to define whether there is a change in exposure to the risk of MSDs (Muskoloskeletal disease) and using fiducial markers for the movement analysis of the operator during the procedure.

DETAILED DESCRIPTION:
Study design: randomized controlled clinical trial. Purpose: Evaluate dentist posture during extraction of third lower molars depending on whether the operator uses the naked eye, surgical loupes or surgical microscope systems. Methods: Data will be analysed through the index RULA (rapid upper limb assesment) to define whether there is a change in exposure to the risk of MSDs (Muskoloskeletal disease).

Posture assessment will be based on 3-D data of the upper body, which can discriminate spatial displacements up to 2mm in translation and 1 degree in rotation.

The surgical intervention will be performed under local anesthesia (mepivacaine 20 mg/ml with adrenaline 1:100000) and by the use of microscope (OPMI Movena S7) or surgical loupes or no magnifying system.

During this session the following data will be collected for the study:

1. Demographic data (baseline)
2. Medical and dental history
3. Parameters related to the lower third molar
4. Radiographic tests
5. Marker operator position
6. Pre- and postoperative photographs

Each patients will be recalled for follow-up visits at 7 days. During this session will be carried out the removal of stitches and data will be recorded as follows:

1. VAS pain and trismus.
2. Number of painkillers taken
3. Control photographs
4. Posse Scala

ELIGIBILITY:
Inclusion Criteria:

* patients elements 38 or 48 in dysodontiasis requiring a complex extraction
* able to sign informed consent

Exclusion Criteria:

* general contraindication to surgical treatment
* pregnancy
* lactation
* age under 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Posture and fatiguing positions | During the surgical procedure (one frame every second during the intervention)
  Specific postural analysis using fiducial markers: a set of markers on the back of a tight T-shirt worn by the dentist during the whole operation will be acquired using a 5 MPixels camera at 2 fps.
  We will place the markers in order to focus our analysis on the following parameter: the neck position with respect to the trunk, the trunk orientation with respect to the vertical axis, the twist and bending of the neck and back, the overall static position duration of the neck and the back.
  The rotation angles of every marker will be extracted and stored for every frame of the recorder video.
Rapid Upper Limb Assessment (RULA) | After the operative performance, an average 15 minutes
  Evaluation tool for ergonomic investigations of workplaces. Values are expressed as RULA scores.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Lodi, PhD, DMD, Principal Investigator — University of Milan
Locations (1):
- University of Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided